CLINICAL TRIAL: NCT02942992
Title: Implementing Resistance Exercise to Reduce Frailty for Older Adult Medicaid Waiver Recipients
Brief Title: Implementing Resistance Exercise to Reduce Frailty for Older Adult
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Margaret Danilovich, Instructor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STU00201777
Record Dates: First submitted 2016-10-04; First posted 2016-10-24 (Estimated); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Usual Care Group
- Intervention (Other): Intervention Group
  Interventions: Behavioral: Resistance exercise

INTERVENTIONS:
Behavioral: Resistance exercise — resistance exercise
  Arms: Intervention

SUMMARY:
To develop an intervention specifically targeted for these clients who have the frailty syndrome. The Investigators propose to develop an exercise intervention that can reduce frailty in older adults to facilitate their ability to age-in-place. The long-term objective of this work is to develop a package of interventions that can be administered within the existing Medicaid Home and Community Based Services (HCBS) Waiver programs. The specific goal of this proposal is to develop a resistance exercise intervention to reduce frailty in older adults receiving long term care services in their home through the Illinois Community Care Program, a HCBS Waiver Program.

ELIGIBILITY:
Inclusion criteria for Home Care Aides:

- Employees of Help at Home, with one eligible client

Inclusion criteria for clients:

* aged 65+ years
* receive HCA services two or more days per week
* English-speaking
* not currently participating in regular exercise as defined as 30 minutes three or more days per week, - - no health problems that contraindicate participation in exercise based on the EASY: Exercise Assessment and Screening for You
* Telephone Interview for Cognitive Status score > 26

Exclusion criteria for HCAs:

- no clients who enroll in the study

Exclusion criteria for clients:

* legally blind, no voluntary extremity movement
* physician does not provide clearance for participation
* classified as non-frail based on the SHARE-FI frailty testing
* Telephone Cognitive Status score < 25.

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 126 (Actual)
Dates: Start 2017-03-30 (Actual); Primary Completion 2017-08-08 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Number of participants with frailty or pre-frailty as assessed by the SHARE-FI | 26 weeks

SECONDARY OUTCOMES:
Scores of self-reported overall health as measured by the PROMIS-global health | 26 weeks
Quadriceps muscle strength as assessed by the 30 second chair rise test | 26 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern Univiersity Department of Physical Therapy and Human Movement Sciences, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Danilovich MK, Diaz L, Ciolinio JD, Corcos DM. Functional resistance activities to impact frailty: A protocol for a randomized controlled trial involving home care aide and frail older adult dyads. Contemp Clin Trials Commun. 2017 May 12;7:28-32. doi: 10.1016/j.conctc.2017.05.006. eCollection 2017 Sep. PMID 29696165